CLINICAL TRIAL: NCT04658537
Title: Advanced Techniques for Single-fraction Palliative Radiotherapy Versus Standard Single Fraction Radiation
Brief Title: Advanced Techniques for Single-fraction Palliative Radiotherapy Versus ASPIRE-single
Acronym: ASPIRE single
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal North Shore Hospital (Other)
Responsible Party: Principal Investigator, Professor Thomas Eade, Radiation Oncologist, Royal North Shore Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASPIRE-single
Record Dates: First submitted 2020-11-24; First posted 2020-12-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Palliative Radiotherapy; Radiotherapy, Intensity-Modulated
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: Non Comparative Randomised Trial
Who Masked: Investigator
Masking Description: Treatment arm will be masked to investigators. Participants will not be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Arm (Active Comparator): 8 Gy / 1 Fraction
  Interventions: Radiation: Radiation Therapy
- Single Fraction Dose Escalation (Experimental): 8Gy Planning Target Volume / 12Gy Clinical Target Volume +/- 14Gy Gross Tumour Volume / 1 fraction
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — Cancer treatment that uses high doses of radiation to kill cancer cells and shrink tumours

SUMMARY:
One third of patients treated in the radiation oncology departments are treated with palliative intent. These patients can be unwell due to their advanced disease and suffering from pain and other symptoms related to metastases. Radiation therapy (RT) has an important role in the symptomatic relief and improvement in the quality of life (QoL) for these patients.The aim of the study is to determine if escalated single fraction palliative radiotherapy using intensity-modulated techniques results in a prolonged duration of benefit for patients otherwise suitable for standard single fraction radiotherapy.

DETAILED DESCRIPTION:
Radiation therapy (RT) has an important role in the symptomatic relief and improvement in the quality of life (QoL) for palliative patients who can be unwell due to their advanced disease and who suffer from pain and other symptoms related to metastases.

A single fraction of 8Gy is considered a standard treatment. In an assessment of health related quality of life (HRQoL) after palliative RT for painful bone metastases, the overall radiotherapy response at 1 week was 45% and by week 2 was 62%. Patients had a significant decrease in pain, insomnia and constipation by 1 month post treatment and an improvement in emotional functioning. When RT is used to control a bleeding tumour, up to 90% of patients will experience haemostasis.

There is however concern that 8 Gy in 1 fraction will not provide a durable response, with up to 20% of patients requiring retreatment to the same site, compared with 8% who receive multiple fraction treatment. Single fraction palliative radiation therapy (SFRT) is therefore an under utilised treatment regimen.

To implement the higher doses with a single fraction, more advanced radiation techniques are required, and there is still equipoise regarding the benefits. With advances in linear accelerator design and software, it is now possible to treat patients with advanced radiation techniques and low resources. Standard clinical pathways including computer optimised planning, remote (virtual) QA of plan delivery and the use of diagnostic imaging for planning are all feasible (under currently in clinical use at Northern Sydney Cancer Centre).

The results from this study will be used to design / proceed to a Randomised Phase III study, if appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic cancer
* Recommended for 8Gy/1# palliative radiation
* Patients with spinal cord compression are eligible for enrolment

Exclusion Criteria:

* Unwilling or unable to give informed consent
* Patients who are recommended multi fraction palliative radiation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-29 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Substantial benefit from palliative radiotherapy | 9 months
  to determine the percentage of patients who achieved a substantial benefit from palliative radiotherapy and have not redeveloped symptoms by 9 months post treatment.

SECONDARY OUTCOMES:
Treatment Wait Time | 1 week
  The time from the date of the initial consultation and radiation therapy consent to the start date of radiation therapy
Radiation Department Time | 1 day
  The time in the radiation oncology department for radiation therapy, from arrival time in the department until the patient is ready for collection at the end of treatment
Radiotherapy Treatment Time | 1 day
  The time that the patient is in the Radiation therapy treatment room, from time of entry to time of exit
Completion Rates of ePRO's in a Palliative Care Cohort | 2 years
  The rate at which baseline and post treatment questionnaires are completed by both patients and primary carers
Comparing Patient and Carer Assessments | 2 years
  Comparing the answers given by patients and carers to determine whether carers can accurately answer on behalf of patients
Radiation Doses to Organs at Risk | 2 years
  The radiation doses delivered to the surrounding organs at risk will be reviewed during and after treatment completion to ensure that they meet predefined OAR constraints Patient and carer reported toxicity from treatment
Patient Reported Outcomes | 24 months
  Electronic questionnaires delivered to the patient pre-treatment and post treatment at 1, 3, 6, 9, 12, 18, and 24 months. Scores will be calculated in accordance with established scoring methods
Carer Reported Outcomes | 24 months
  Electronic questionnaires delivered to the patient's primary carer pre-treatment and post treatment at 1, 3, 6, 9, 12, 18, and 24 months. Scores will be calculated in accordance with established scoring methods
Efficacy of treatment | 2 years
  this will be determined by re-treatment rates of irradiated sites, symptom control and recurrence
Overall Survival | 2 years
  This will be defined as the time to death measured from the day of randomisation.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Eade, Principal Investigator — Department of Radiation Oncology, Northern Sydney Cancer Centre, Royal North Shore Hospital
Locations (1):
- Royal North Shore Hospital, Saint Leonards, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
The results of this trial will be published in a peer reviewed journal. Target journals for publication of this trial include, International Journal of Radiation Oncology Biology Physics

REFERENCES:
- [Background] Wu JS, Wong R, Johnston M, Bezjak A, Whelan T; Cancer Care Ontario Practice Guidelines Initiative Supportive Care Group. Meta-analysis of dose-fractionation radiotherapy trials for the palliation of painful bone metastases. Int J Radiat Oncol Biol Phys. 2003 Mar 1;55(3):594-605. doi: 10.1016/s0360-3016(02)04147-0. PMID 12573746
- [Background] Rich SE, Chow R, Raman S, Liang Zeng K, Lutz S, Lam H, Silva MF, Chow E. Update of the systematic review of palliative radiation therapy fractionation for bone metastases. Radiother Oncol. 2018 Mar;126(3):547-557. doi: 10.1016/j.radonc.2018.01.003. Epub 2018 Feb 1. PMID 29397209
- [Background] Caissie A, Zeng L, Nguyen J, Zhang L, Jon F, Dennis K, Holden L, Culleton S, Koo K, Tsao M, Barnes E, Danjoux C, Sahgal A, Simmons C, Chow E. Assessment of health-related quality of life with the European Organization for Research and Treatment of Cancer QLQ-C15-PAL after palliative radiotherapy of bone metastases. Clin Oncol (R Coll Radiol). 2012 Mar;24(2):125-33. doi: 10.1016/j.clon.2011.08.008. Epub 2011 Sep 13. PMID 21917431
- [Background] Sapienza LG, Ning MS, Jhingran A, Lin LL, Leao CR, da Silva BB, Pellizzon ACA, Gomes MJL, Baiocchi G. Short-course palliative radiation therapy leads to excellent bleeding control: A single centre retrospective study. Clin Transl Radiat Oncol. 2018 Nov 22;14:40-46. doi: 10.1016/j.ctro.2018.11.007. eCollection 2019 Jan. PMID 30555940
- [Background] Wu SY, Singer L, Boreta L, Garcia MA, Fogh SE, Braunstein SE. Palliative radiotherapy near the end of life. BMC Palliat Care. 2019 Mar 23;18(1):29. doi: 10.1186/s12904-019-0415-8. PMID 30904024
- [Background] Schuler T, Back M, Hruby G, Carroll S, Jayamanne D, Kneebone A, Stevens M, Lamoury G, Morgia M, Wong S, Grimberg K, Roderick S, Booth J, Eade T. Introducing Computed Tomography Simulation-Free and Electronic Patient-Reported Outcomes-Monitored Palliative Radiation Therapy into Routine Care: Clinical Outcomes and Implementation Experience. Adv Radiat Oncol. 2020 Dec 3;6(2):100632. doi: 10.1016/j.adro.2020.100632. eCollection 2021 Mar-Apr. PMID 33851063
- [Background] Nguyen QN, Chun SG, Chow E, Komaki R, Liao Z, Zacharia R, Szeto BK, Welsh JW, Hahn SM, Fuller CD, Moon BS, Bird JE, Satcher R, Lin PP, Jeter M, O'Reilly MS, Lewis VO. Single-Fraction Stereotactic vs Conventional Multifraction Radiotherapy for Pain Relief in Patients With Predominantly Nonspine Bone Metastases: A Randomized Phase 2 Trial. JAMA Oncol. 2019 Jun 1;5(6):872-878. doi: 10.1001/jamaoncol.2019.0192. PMID 31021390
- [Background] Ryu S, Deshmukh S, Timmerman RD, Movsas B, Gerszten PC, Yin FF, et al. Radiosurgery Compared To External Beam Radiotherapy for Localized Spine Metastasis: Phase III Results of NRG Oncology/RTOG 0631. International Journal of Radiation Oncology • Biology • Physics. 2019;105(1):S2-S3.
- [Background] Ong WL, Foroudi F, Milne RL, Millar JL. Variation in the Use of Single- Versus Multifraction Palliative Radiation Therapy for Bone Metastases in Australia. Int J Radiat Oncol Biol Phys. 2020 Jan 1;106(1):61-66. doi: 10.1016/j.ijrobp.2019.08.061. Epub 2019 Sep 7. PMID 31505246
- [Background] Roos DE, Turner SL, O'Brien PC, Smith JG, Spry NA, Burmeister BH, Hoskin PJ, Ball DL; Trans-Tasman Radiation Oncology Group, TROG 96.05. Randomized trial of 8 Gy in 1 versus 20 Gy in 5 fractions of radiotherapy for neuropathic pain due to bone metastases (Trans-Tasman Radiation Oncology Group, TROG 96.05). Radiother Oncol. 2005 Apr;75(1):54-63. doi: 10.1016/j.radonc.2004.09.017. Epub 2004 Oct 28. PMID 15878101
- [Background] Maranzano E, Bellavita R, Rossi R, De Angelis V, Frattegiani A, Bagnoli R, Mignogna M, Beneventi S, Lupattelli M, Ponticelli P, Biti GP, Latini P. Short-course versus split-course radiotherapy in metastatic spinal cord compression: results of a phase III, randomized, multicenter trial. J Clin Oncol. 2005 May 20;23(15):3358-65. doi: 10.1200/JCO.2005.08.193. Epub 2005 Feb 28. PMID 15738534
- [Background] Maranzano E, Trippa F, Casale M, Costantini S, Lupattelli M, Bellavita R, Marafioti L, Pergolizzi S, Santacaterina A, Mignogna M, Silvano G, Fusco V. 8Gy single-dose radiotherapy is effective in metastatic spinal cord compression: results of a phase III randomized multicentre Italian trial. Radiother Oncol. 2009 Nov;93(2):174-9. doi: 10.1016/j.radonc.2009.05.012. Epub 2009 Jun 10. PMID 19520448
- [Background] Lee KA, Dunne M, Small C, Kelly PJ, McArdle O, O'Sullivan J, Hacking D, Pomeroy M, Armstrong J, Moriarty M, Clayton-Lea A, Parker I, Collins CD, Thirion P. (ICORG 05-03): prospective randomized non-inferiority phase III trial comparing two radiation schedules in malignant spinal cord compression (not proceeding with surgical decompression); the quality of life analysis. Acta Oncol. 2018 Jul;57(7):965-972. doi: 10.1080/0284186X.2018.1433320. Epub 2018 Feb 8. PMID 29419331
- [Background] Job M, Holt T, Bernard A. Reducing radiotherapy waiting times for palliative patients: The role of the Advanced Practice Radiation Therapist. J Med Radiat Sci. 2017 Dec;64(4):274-280. doi: 10.1002/jmrs.243. Epub 2017 Aug 29. PMID 28851033
- [Background] Thavarajah N, Wong K, Zhang L, Bedard G, Wong E, Tsao M, Danjoux C, Barnes E, Sahgal A, Dennis K, Holden L, Lauzon N, Chow E. Continued success in providing timely palliative radiation therapy at the Rapid Response Radiotherapy Program: a review of 2008-2012. Curr Oncol. 2013 Jun;20(3):e206-11. doi: 10.3747/co.20.1342. PMID 23737690
- [Background] Wong S, Roderick S, Atyeo JW, Grimberg K, Porter B, Booth J, et al. Improving the Palliative Patient Journey in Radiation Oncology. International Journal of Radiation Oncology • Biology • Physics. 2019;105(1):S49.
- [Background] Sandler KA, Mitchell SA, Basch E, Raldow AC, Steinberg ML, Sharif J, Cook RR, Kupelian PA, McCloskey SA. Content Validity of Anatomic Site-Specific Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) Item Sets for Assessment of Acute Symptomatic Toxicities in Radiation Oncology. Int J Radiat Oncol Biol Phys. 2018 Sep 1;102(1):44-52. doi: 10.1016/j.ijrobp.2018.04.048. Epub 2018 Jun 5. PMID 30102201
- [Background] Brunelli C, Zecca E, Martini C, Campa T, Fagnoni E, Bagnasco M, Lanata L, Caraceni A. Comparison of numerical and verbal rating scales to measure pain exacerbations in patients with chronic cancer pain. Health Qual Life Outcomes. 2010 Apr 22;8:42. doi: 10.1186/1477-7525-8-42. PMID 20412579
- See also: Varian. Varian Adaptive Therapy Ethos. — https://www.varian.com/en-au/products/adaptive-therapy/ethos